CLINICAL TRIAL: NCT04483245
Title: Platelet Activation by a Collagen Analogue in Hemorrhagic Situations
Acronym: CAPTURE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DE MAISTRE 2019
Record Dates: First submitted 2020-07-17; First posted 2020-07-23 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Collagen Analog; Platelet Activation; Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- controls: persons free of hemorrhage or haemostasis disorder
  Interventions: Biological: Blood sampling
- Haemorrhagic: Acute hemorrhagic patient
  Interventions: Biological: Blood sampling
- ECMO: ECMO surgery patient with hemorrhagic complication
  Interventions: Biological: Blood sampling
- polytrauma
  Interventions: Biological: Blood sampling
- Platelet disorder: Patient with an identified platelet disorder or treated with antiplatelet agents
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — Blood sampling

SUMMARY:
Dijon University Hospital and the Dijon-based NVH Medicinal Company have developed a recombinant mini-collagen NVH020B with platelet and Willebrand factor binding activity. Its small size and granular, non-fibrillar presentation make it suitable for use as an injectable hemostat in patients with a hemorrhage or other emergency under antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* - person who has given their non-opposition to inclusion
* adult
* Healthy volunteers or controls (patients seen in consultation, without history of hemmorhage, etc.).

or

* patients with acute bleeding: polytraumatized, or hemorrhage or intracerebral haemorrhage, or bleeding complications at the end surgery (in particular cardiac surgery with ECMO) or
* patients with antiplatelet therapy or
* patients with thrombocytopenia/thrombopathy

Exclusion Criteria:

* protected adults (curatorship, guardianship)
* person deprived of their liberty by judicial or administrative decision
* pregnant, parturient or breastfeeding woman
* person unable to express their non-opposition
* platelet transfusion on initial management

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients coming for a consultation at the Resouce Centre for Haemorrhagic Diseases and Coagulopathies in the Internal Medicine and Haematology Department. Patients admitted to the Emergency Department, and patients admitted to the operating theatre by the Surgical Intensive Care Unit, the Neurovascular Emergency Department, or the Neurosurgery Department.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
The expression of P-selectin and activated GPIIb/IIIa (PAC1) at the surface of platelets in flow cytometry in response to NVH020B. | Through study completion, an average of 1 year
  These 2 markers are absent on the surface of resting platelets. The expression of these 2 markers will make it possible to evaluate the role of the mini-collagen as an activator.

SECONDARY OUTCOMES:
Platelet aggregation rate in response to NVH020B | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France